CLINICAL TRIAL: NCT05353361
Title: A Phase Ib/II Multicenter, Open-Label Clinical Trial of SHR-A1811 Injection in Combination With Pyrotinib or Pertuzumab or Adebrelimab or Paclitaxel for Injection (Albumin Bound) in Breast Cancer
Brief Title: A Phase Ib/II Study of SHR-A1811 Injection in Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-II-202
Record Dates: First submitted 2022-04-19; First posted 2022-04-29 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This study is a multicenter, open-label, dose exploration and efficacy expansion phase Ib / II study. The first stage is the dose exploration phase, which uses the 3 + 3 escalation design; The second stage is the curative effect expansion phase.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SHR-A1811combined Pyrotinib (Experimental)
  Interventions: Drug: SHR-A1811：Pyrotinib
- SHR-A1811Combined Pertuzumab (Experimental)
  Interventions: Drug: SHR-A1811；Pertuzumab
- SHR-A1811Combined Adebrelimab (Experimental)
  Interventions: Drug: SHR-A1811；Adebrelimab
- SHR-A1811Combined Albumin-bound Paclitaxel (Experimental)
  Interventions: Drug: SHR-A1811；Albumin paclitaxel

INTERVENTIONS:
Drug: SHR-A1811：Pyrotinib — SHR-A1811：Lyophilized powder injection, 100mg / bottle, intravenous drip Pyrotinib：Tablet, 160mg / tablet, 80mg / tablet, oral
  Arms: SHR-A1811combined Pyrotinib
Drug: SHR-A1811；Pertuzumab — SHR-A1811：Lyophilized powder injection, 100mg / bottle, intravenous drip Pertuzumab：Injection, 420 Mg (14 ml) / bottle, intravenous drip
  Arms: SHR-A1811Combined Pertuzumab
Drug: SHR-A1811；Adebrelimab — SHR-A1811：Lyophilized powder injection, 100mg / bottle, intravenous drip Adebrelimab：Injection, 12ml: 0.6g/bottle, intravenous drip
  Arms: SHR-A1811Combined Adebrelimab
Drug: SHR-A1811；Albumin paclitaxel — SHR-A1811：Lyophilized powder injection, 100mg / bottle, intravenous drip Albumin paclitaxel：Injection, 100mg / box, intravenous drip
  Arms: SHR-A1811Combined Albumin-bound Paclitaxel

SUMMARY:
To evaluate the safety, tolerability and efficacy of SHR-A1811 in combination with pyrotinib or pertuzumab or adebrelimab or albumin-bound paclitaxel in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 to 75 (inclusive)
2. Breast cancer confirmed by histology or cytology.
3. ECOG score is 0 or 1
4. An expected survival of ≥ 12 weeks
5. At least one measurable lesion according to RECIST v1.1 criteria
6. Have adequate renal and hepatic function
7. Patients voluntarily joined the study and signed informed consent

Exclusion Criteria:

1. Have other malignancies within the past 5 years
2. Active central nervous system metastasis without surgery or radiotherapy
3. Presence with uncontrollable third space effusion
4. Have undergone other anti-tumor treatment within 4 weeks before the first dose
5. Immunosuppressant or systemic hormone therapy was used within 2 weeks prior to the first dose
6. Any active autoimmune disease or a history of autoimmune disease
7. A history of immune deficiency
8. Clinically significant cardiovascular disorders
9. Clinically significant history of lung disease
10. The toxicity from previous anti-tumor treatment has not recovered to ≤ grade I
11. Known hereditary or acquired bleeding tendency
12. Active hepatitis and liver cirrhosis
13. Presence of other serious physical or mental diseases or laboratory abnormalities

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
DLT（Phase I (dose exploration phase) ） | 21 days after the first administration of each subject
AE（Phase I (dose exploration phase) ） | from Day1 to 40 or 90 days after last dose
Incidence and severity of serious adverse events (SAE)（Phase I (dose exploration phase) ） | from Day1 to 40 or 90 days after last dose
Objective response rate（Phase II (efficacy expansion phase)） | Two years after the last subject was enrolled in the group

SECONDARY OUTCOMES:
PK parameter: Cmin of SHR-A1811（Phase I secondary endpoint） | through study completion, an average of 2 years
PK parameter: Cmax of SHR-A1811（Phase I secondary endpoint） | through study completion, an average of 2 years
PK parameter: AUC0-t of SHR-A1811（Phase I secondary endpoint） | through study completion, an average of 2 years
PK parameter: Cmin of Pyrotinib（Phase I secondary endpoint） | through study completion, an average of 2 years
PK parameter: C4h of Pyrotinib（Phase I secondary endpoint） | through study completion, an average of 2 years
PK parameter: Cmin of Adebrelimab（Phase I secondary endpoint） | through study completion, an average of 2 years
Immunogenicity of SHR-A1811（Phase I secondary endpoint） | through study completion, an average of 2 years
Immunogenicity of Adebrelimab（Phase I secondary endpoint） | through study completion, an average of 2 years
Objective Response Rate（Phase I secondary endpoint） | from first dose to disease progression or death, whichever comes first, up to 3 years
Duration of response（Phase I secondary endpoint） | from first dose to disease progression or death, whichever comes first, up to 3 years
Progression Free Survival（Phase I secondary endpoint） | from first dose to disease progression or death, whichever comes first, up to 3 years
AE（Phase II secondary study endpoint） | from Day1 to 40 or 90 days after last dose
Incidence and severity of serious adverse events (SAE)（Phase II secondary study endpoint） | from Day1 to 40 or 90 days after last dose
PK parameter: Cmin, Cmax, and AUC0-t of SHR-A1811（Phase II secondary study endpoint） | through study completion, an average of 2 years
PK parameter: Cmin, C4h of Pyrotinib:（Phase II secondary study endpoint） | through study completion, an average of 2 years
PK parameter: Cmin of Adebrelimab（Phase II secondary study endpoint） | through study completion, an average of 2 years
Immunogenicity of SHR-A1811（Phase II secondary study endpoint） | through study completion, an average of 2 years
Immunogenicity of Adebrelimab（Phase II secondary study endpoint） | through study completion, an average of 2 years
Duration of response（Phase II secondary study endpoint） | from first dose to disease progression or death, whichever comes first, up to 3 years
Progression Free Survival（Phase II secondary study endpoint） | from first dose to disease progression, or death, whichever comes first, up to 3 years
Event-Free Survival Rate（Phase II secondary study endpoint） | from first dose to disease progression, disease recurrence, or death, whichever comes first, up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Provincial People's Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided